CLINICAL TRIAL: NCT00941863
Title: Phase I Study to Determine the Safety, Maximum Tolerated Dose, PK of BAY43-9006 in Repeated Cycles of 18 Days On/3 Days Off in Combination With Paclitaxel and Carboplatin Chemotherapy in Patients With Advanced, Refractory Solid Tumors
Brief Title: Study to Determine the Safety, Maximum Tolerated Dose, Pharmacokinetics of Sorafenib (BAY43-9006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100375
Record Dates: First submitted 2009-06-12; First posted 2009-07-20 (Estimated); Results first posted 2010-10-08 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Carcinoma
Keywords: Sorafenib; Advanced Solid Tumors; Maximum tolerated dose; Carboplatin and paclitaxel chemotherapy combination
MeSH Terms: conditions — Carcinoma | interventions — Sorafenib; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sorafenib 100 mg (50-mg tablet) (Experimental): Dose-escalation cohort 1: Sorafenib (Nexavar, BAY43-9006) 100 mg twice daily (50-mg tablet). Treatment were planned until primary completion date (PCD).
  Interventions: Drug: Sorafenib 100 mg (50-mg tablet)
- Sorafenib 200 mg (50-mg tablet) (Experimental): Dose-escalation cohort 2: Sorafenib (Nexavar, BAY43-9006) 200 mg twice daily (50-mg tablet). Treatment were planned until primary completion date (PCD).
  Interventions: Drug: Sorafenib 200 mg (50-mg tablet)
- Sorafenib 400 mg (50-mg tablet) (Experimental): Dose-escalation cohort 3: Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (50-mg tablet). Treatment were planned until primary completion date (PCD).
  Interventions: Drug: Sorafenib 400 mg (50-mg tablet)
- Sorafenib 400 mg (200-mg tablet) (Experimental): Dose-escalation cohort 4: Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (200-mg tablet). Treatment were planned until primary completion date (PCD).
  Interventions: Drug: Sorafenib 400 mg (200-mg tablet)
- Sorafenib 400 mg (Expansion) (Experimental): Dose-expansion cohort: Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (200-mg tablet) expansion. Treatment were planned until primary completion date (PCD). 25 of 119 participants from the Expansion Phase, were still on the treatment as of 31 May 2005. Of these, 6 subjects were continuing to receive sorafenib in combination with carboplatin and/or paclitaxel and 19 subjects were receiving single-agent sorafenib until 18 Sep 2008.
  Interventions: Drug: Sorafenib 400 mg (Expansion)

INTERVENTIONS:
Drug: Sorafenib 100 mg (50-mg tablet) — Sorafenib (Nexavar, BAY43-9006) 100 mg twice daily (50-mg tablet)
  Arms: Sorafenib 100 mg (50-mg tablet)
Drug: Sorafenib 200 mg (50-mg tablet) — Sorafenib (Nexavar, BAY43-9006) 200 mg twice daily (50-mg tablet)
  Arms: Sorafenib 200 mg (50-mg tablet)
Drug: Sorafenib 400 mg (50-mg tablet) — Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (50-mg tablet)
  Arms: Sorafenib 400 mg (50-mg tablet)
Drug: Sorafenib 400 mg (200-mg tablet) — Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (200-mg tablet)
  Arms: Sorafenib 400 mg (200-mg tablet)
Drug: Sorafenib 400 mg (Expansion) — Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (200-mg tablet) expansion
  Arms: Sorafenib 400 mg (Expansion)

SUMMARY:
The primary objective of the study was to define the safety profile and maximum tolerated dose (MTD) of sorafenib tablets in combination with carboplatin and paclitaxel chemotherapy in patients with advanced, refractory solid tumors.

The secondary objectives were evaluation of pharmacokinetics (PK) and tumor response of these patients being treated with sorafenib in combination with paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors
* Evaluable disease
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Life expectancy minimum 12 weeks

Exclusion Criteria:

* Congestive heart failure
* Serious arrhythmias
* Coronary artery disease (CAD) or ischemia
* HIV (human immunodeficiency virus)
* Hepatitis B or C
* Serious active infection
* Metastatic brain or meningeal tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2002-07; Primary Completion 2005-05 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- United States (3):
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 centers in the US: the University of Wisconsin, the University of Pennsylvania, and Vanderbilt University. Enrollment began 01 Jul 2002.
Pre-assignment Details: Expansion in this context is an increase in the number of patients exposed to the recommended dose for this combination. The purpose of the increase was also to test efficacy signals in Metastatic Melanoma (MM).
Groups:
- Sorafenib 100 mg (50-mg Tablet): Dose-escalation cohort 1: Sorafenib (Nexavar, BAY43-9006) 100 mg twice daily (50-mg tablet)
- Sorafenib 200 mg (50-mg Tablet): Dose-escalation cohort 2: Sorafenib (Nexavar, BAY43-9006) 200 mg twice daily (50-mg tablet)
- Sorafenib 400 mg (50-mg Tablet): Dose-escalation cohort 3: Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (50-mg tablet)
- Sorafenib 400 mg (200-mg Tablet): Dose-escalation cohort 4: Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (200-mg tablet)
- Sorafenib 400 mg (Expansion): Dose-expansion cohort: Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (200-mg tablet) expansion
Period: Until Primary Completion Date (PCD)
Arm/Group | Sorafenib 100 mg (50-mg Tablet) | Sorafenib 200 mg (50-mg Tablet) | Sorafenib 400 mg (50-mg Tablet) | Sorafenib 400 mg (200-mg Tablet) | Sorafenib 400 mg (Expansion)
Started | 7 | 3 | 12 | 17 | 119
Maximum Tolerated Dose | 7 | 3 | 12 | 17 | 94
Completed | 0 | 0 | 0 | 0 | 25
Not Completed | 7 | 3 | 12 | 17 | 94
Not completed — Adverse Event | 1 | 2 | 2 | 1 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 8
Not completed — Death | 0 | 0 | 1 | 2 | 7
Not completed — Disease progression | 6 | 1 | 8 | 14 | 73
Period: Continued After PCD
Arm/Group | Sorafenib 100 mg (50-mg Tablet) | Sorafenib 200 mg (50-mg Tablet) | Sorafenib 400 mg (50-mg Tablet) | Sorafenib 400 mg (200-mg Tablet) | Sorafenib 400 mg (Expansion)
Started | 0 | 0 | 0 | 0 | 25 (25 of 119 participants from the Expansion Phase, were still on the treatment as of 31 May 2005.)
Completed | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 19
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Disease progression, recurrence, relapse | 0 | 0 | 0 | 0 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib 100 mg (50-mg Tablet) | Sorafenib 200 mg (50-mg Tablet) | Sorafenib 400 mg (50-mg Tablet) | Sorafenib 400 mg (200-mg Tablet) | Sorafenib 400 mg (Expansion) | Total
Number analyzed (Participants) | 7 | 3 | 12 | 17 | 119 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (17.9) | 52.0 (12.0) | 52.0 (14.4) | 52.8 (10.5) | 52.8 (12.6) | 52.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 7 | 54 | 67
  Male | 5 | 2 | 9 | 10 | 65 | 91
Race/Ethnicity, Customized [Number; unit: participants]
  white | 6 | 3 | 12 | 16 | 113 | 150
  black | 0 | 0 | 0 | 0 | 2 | 2
  asian | 0 | 0 | 0 | 1 | 2 | 3
  hispanic | 1 | 0 | 0 | 0 | 2 | 3
Site of primary lesion [Number; unit: participants] — Tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
  participants
    Colon | 1 | 0 | 1 | 2 | 1 | 5
    Malignant Melanoma | 3 | 1 | 10 | 10 | 81 | 105
    Non Small Cell Lung | 1 | 0 | 1 | 2 | 11 | 15
    Ovarian | 0 | 0 | 0 | 0 | 3 | 3
    Renal | 0 | 1 | 0 | 1 | 21 | 23
    Other | 2 | 1 | 0 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Sorafenib in Combination With Paclitaxel and Carboplatin
Description: MTD was determined by testing increasing doses up to 400 mg twice daily (bid) on dose escalation cohorts 1 to 3 with 3 patients each. MTD reflects highest dose of drug that did not cause an unacceptable side effect (= Dose Limiting Toxicity (DLT) in more than 30% of patients; e.g., hematologic toxicities like Common Toxicity Criteria (CTC) Grade 4 Neutropenia in specific conditions, platelets < 25,000 cells/mL; specific non-hematologic/biochemical toxicities CTC Grade 3 or 4; additionally, any toxicity considered by the investigator severe enough was designated a DLT); CTC Version 2 were used.
Time Frame: 21 days
Population: All subjects who received at least 1 dose of any study drug treatment were included in the Intent-To-Treat/safety populations. Efficacy parameters of time to death, time to progression, and response rate (confirmed partial response [PR] plus complete response [CR]) were determined for this population.
Measure: Number; unit: mg
Groups:
- Sorafenib, Dose Escalation 100 mg Bid, 200 mg Bid, 400 mg Bid: All participants of escalation cohorts 1, 2, 3 and 4. (Sorafenib, dose escalation 100 mg bid [twice daily], 200 mg bid, 400 mg bid including 50 tablet and 200 tablet)
Arm/Group | Sorafenib, Dose Escalation 100 mg Bid, 200 mg Bid, 400 mg Bid
Number analyzed (Participants) | 39
mg | 400

2. Primary Outcome: Participants With Hematological and Biochemical Toxicities
Description: Participants are considered at risk for toxicity if participants had a lab measurement for the toxicity >= National Cancer Institute Common Toxicity Criteria (NCI CTC) Grade 3 as defined by the NCI CTC version 2; SGOT: Serum Glutamic-Oxaloacetic Transaminase, SGPT: Serum Glutamic-Pyruvic Transaminase, AST: Aspartate Aminotransferase, ALT: Alanine Aminotransferase.
Time Frame: Start of treatment until death or within 14 days last study drug intake
Population: The Intent-To-Treat (ITT) population included subjects who received at least one dose of sorafenib or chemotherapy and had at least one post baseline assessment. Efficacy analyses were performed on the ITT population.
Measure: Number; unit: Participants
Groups:
- Sorafenib 400 mg (Expansion, Treatment Until PCD): Dose-expansion cohort: Sorafenib (Nexavar, BAY43-9006) 400 mg twice daily (200-mg tablet) expansion
- Sorafenib 400 mg (Expansion, Treatment Continued After PCD): 25 of 119 participants from the Expansion Phase, were still on the treatment as of 31 May 2005. Of these, 6 subjects were continuing to receive sorafenib in combination with carboplatin and/or paclitaxel and 19 subjects were receiving single-agent sorafenib. The responses reported in these participants were from start of treatment until 18 Sep 2008.
Arm/Group | Sorafenib 100 mg (50-mg Tablet) | Sorafenib 200 mg (50-mg Tablet) | Sorafenib 400 mg (50-mg Tablet) | Sorafenib 400 mg (200-mg Tablet) | Sorafenib 400 mg (Expansion, Treatment Until PCD) | Sorafenib 400 mg (Expansion, Treatment Continued After PCD)
Number analyzed (Participants) | 7 | 3 | 12 | 17 | 119 | 25
Participants
  Hemoglobin >= NCI CTC Grade 3 | 1 | 0 | 2 | 5 | 28 | 6
  Leukocytes >= NCI CTC Grade 3 | 7 | 1 | 10 | 14 | 95 | 17
  Lymphopenia >= NCI CTC Grade 3 | 5 | 1 | 5 | 11 | 99 | 4
  Neutrophils/ Granulocytes >= NCI CTC Grade 3 | 4 | 2 | 6 | 10 | 87 | 14
  Platelets >= NCI CTC Grade 3 | 1 | 3 | 6 | 8 | 62 | 9
  Bilirubin >= NCI CTC Grade 3 | 0 | 0 | 0 | 0 | 2 | 1
  SGOT (AST) >= NCI CTC Grade 3 | 0 | 0 | 0 | 0 | 5 | 1
  SGPT (ALT) >= NCI CTC Grade 3 | 0 | 0 | 0 | 0 | 5 | 2
  Hypophosphatemia >= NCI CTC Grade 3 | 3 | 1 | 2 | 8 | 52 | 12

3. Secondary Outcome: Tumor Response
Description: Tumor Response (= Best Overall Response) of a subject was defined as the best tumor response (confirmed Complete Response (CR), confirmed Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)) observed during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR was defined as disappearance of tumor lesions, PR was defined as a decrease of at least 30% in the sum of tumor lesion sizes, SD was defined as steady state of disease, PD was defined as an increase of at least 20% in the sum of tumor lesions sizes.
Time Frame: From start of treatment until progression or death occurs assessed every 6 weeks.
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Sorafenib 100 mg (50-mg Tablet) | Sorafenib 200 mg (50-mg Tablet) | Sorafenib 400 mg (50-mg Tablet) | Sorafenib 400 mg (200-mg Tablet) | Sorafenib 400 mg (Expansion, Treatment Until PCD) | Sorafenib 400 mg (Expansion, Treatment Continued After PCD)
Number analyzed (Participants) | 7 | 3 | 12 | 17 | 119 | 25
Participants
  Complete Response (CR) | 0 | 0 | 0 | 1 | 0 | 1
  Partial Response (PR) | 1 | 1 | 4 | 3 | 28 | 12
  Stable Disease (SD) | 4 | 1 | 4 | 10 | 73 | 12
  Progressive Disease (PD) | 2 | 0 | 1 | 2 | 6 | 0
  Not Assessable | 0 | 1 | 3 | 1 | 12 | 0

4. Secondary Outcome: Area Under the Curve From Time 0 to 12 Hours Post-dose (AUC 0-12) Start From Day 2 of Cycle 1
Description: The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. A plot of concentration vs time after dosing is created, and the area under this curve is calculated by standard methods (eg, trapezoidal rule) to provide a measure of how much drug was in the bloodstream following dosing.
Time Frame: At day 2 in study
Population: subjects with valid pharmacokinetics (PK) profiles
Measure: Geometric Mean (Standard Deviation); unit: mg*h/L
Groups:
- Sorafenib 400 mg (Excluding Expansion): Dose-escalation cohorts 3 and 4
Arm/Group | Sorafenib 400 mg (Excluding Expansion)
Number analyzed (Participants) | 25
mg*h/L | 17.5 (2.16)

5. Secondary Outcome: Maximum Concentration (CMAX) Start From Day 2 of Cycle 1
Description: Cmax refers to the highest plasma concentration of drug reached after dosing. It is obtained by collecting a series of blood samples after dosing, and analyzing them for drug content by a sensitive and specific analytical method. The highest measured concentration is referred to as the Cmax.
Time Frame: At day 2 in study
Population: subjects with valid PK profiles
Measure: Geometric Mean (Standard Deviation); unit: mg/L
Arm/Group | Sorafenib 400 mg (Excluding Expansion)
Number analyzed (Participants) | 25
mg/L | 3.36 (1.79)

6. Secondary Outcome: Time of Maximum Concentration (TMAX) Start From Day 2 of Cycle 1
Description: Tmax refers to the time after dosing when a drug attains its maximum concentration in the blood. It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content. The time corresponding to the highest measurable concentration (Cmax) is referred to as Tmax.
Time Frame: At day 2 in study
Population: subjects with valid PK profiles
Measure: Median (Full Range); unit: hours
Arm/Group | Sorafenib 400 mg (Excluding Expansion)
Number analyzed (Participants) | 25
hours | 24.5 [3 to 36.08]

7. Other Pre Specified Outcome: Serious Adverse Events
Description: The responses reported in these participants were from start of treatment until 18 Sep 2008.
Time Frame: From start of treatment until 18 Sep 2008, up to 6 years
Population: 25 of 119 participants from the Expansion Phase, were still on the treatment as of 31 May 2005. Of these, 6 subjects were continuing to receive sorafenib in combination with carboplatin and/or paclitaxel and 19 subjects were receiving single-agent sorafenib.
Measure: Number; unit: Participants
Arm/Group | Sorafenib 400 mg (Expansion, Treatment Continued After PCD)
Number analyzed (Participants) | 25
Participants
  Hemoglobin | 1
  Cardiovascular/Arrhythmia-Other | 1
  Supraventricular Arrhythmias | 3
  Cardiac-Ischemia/Infarction | 2
  Thrombosis/Embolism | 1
  Constitutional Symptoms-Other | 1
  Fatigue | 1
  Fever | 3
  Dermatology/Skin-Other | 1
  Gastrointestinal-Other | 1
  Nausea | 1
  Vomiting | 1
  Hematuria | 1
  Hemoptysis | 1
  Hemorrhage-Other | 1
  Febrile Neutropenia | 2
  Infection Without Neutropenia | 2
  Infection/Febrile Neutropenia-Other | 1
  Hyperglycemia | 1
  Hypoglycemia | 1
  Hypokalemia | 1
  Depressed Level Of Consciousness | 1
  Syncope | 2
  Chest Pain (NonCardiac/NonPleuritic) | 2
  Pain-Other | 1
  Pleural Effusion (Non-Malignant) | 1
  Pneumonitis/Pulmonary Infiltrates | 1
  Renal/Genitourinary-Other | 1

8. Other Pre Specified Outcome: Other Adverse Events
Description: Frequency Threshold for reporting Other Adverse Events: 5%. The responses reported in these participants were from start of treatment until 18 Sep 2008.
Time Frame: From start of treatment until 18 Sep 2008, up to 6 years
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Sorafenib 400 mg (Expansion, Treatment Continued After PCD)
Number analyzed (Participants) | 25
Participants
  Allergic Reaction/Hyper-Sensitivity | 5
  Allergic Rhinitis | 7
  Allergy/ Immunology-Other | 4
  Auditory/Hearing-Other | 2
  Hemoglobin | 14
  Leukocytes | 11
  Neutrophils/Granulocytes | 19
  Platelets | 15
  Cardiovascular/General-Other | 2
  Edema | 6
  Hypertension | 6
  Constitutional Symptoms-Other | 8
  Fatigue | 22
  Fever | 6
  Rigors, Chills | 3
  Sweating (Diaphoresis) | 2
  Weight Loss | 10
  Alopecia | 16
  Dermatology/Skin-Other | 15
  Dry Skin | 5
  Flushing | 3
  Hand-Foot Skin Reaction | 15
  Injection Site Reaction | 3
  Pruritus | 5
  Rash/Desquamation | 20
  Wound-Infectious | 3
  Wound-Non-Infectious | 3
  Anorexia | 14
  Constipation | 7
  Dehydration | 4
  Diarrhea | 18
  Dyspepsia/Heartburn | 5
  Dysphagia,Esophagitis,Odynophagia | 4
  Gastrointestinal-Other | 6
  Nausea | 16
  Stomatitis/Pharyngitis | 9
  Taste Disturbance (Dysgeusia) | 5
  Vomiting | 11
  Epistaxis | 7
  Hemorrhage-Other | 6
  Alkaline Phosphatase | 2
  Bilirubin | 2
  Hypoalbuminemia | 2
  Infection With Unknown Anc | 5
  Infection Without Neutropenia | 14
  Hyperglycemia | 5
  Hypokalemia | 4
  Hypomagnesemia | 8
  Hyponatremia | 3
  Hypophosphatemia | 4
  Arthritis | 2
  Musculoskeletal-Other | 8
  Confusion | 2
  Dizziness/Lightheadedness | 2
  Insomnia | 7
  Memory Loss | 2
  Mood Alteration-Anxiety, Agitation | 5
  Mood Alteration-Depression | 7
  Neurology-Other | 2
  Neuropathy-Motor | 8
  Neuropathy-Sensory | 19
  Vertigo | 2
  Ocular/Visual-Other | 2
  Vision, Blurred Vision | 3
  Abdominal Pain Or Cramping | 6
  Arthralgia (Joint Pain) | 13
  Bone Pain | 8
  Chest Pain (NonCardiac/NonPleuritic) | 5
  Headache | 8
  Myalgia (Muscle Pain) | 16
  Pain-Other | 10
  Tumor Pain | 3
  Cough | 11
  Dyspnea (Shortness Of Breath) | 13
  Pneumonitis/Pulmonary Infiltrates | 2
  Voice Changes/Stridor/Larynx | 3

ADVERSE EVENTS:
Time Frame: Time frame for expansion group is from start of treatment until April 2008, up to 6 years.
Description: Acronyms in Adverse Event Section:
  White Blood Cell (WBC) Absolute Neutrophil Count (ANC) Absolute Granulocyte Count (AGC) Alanine Transaminase (ALT) Aspartate Transaminase (AST) Grade (GR) Gastrointestinal (GI) Central Nervous System (CNS) Fibrillation/Flutter (FIB/FLUTT) Neutropenia (Neu) documented (doc)
Arm/Group | Sorafenib 100 mg (50-mg Tablet) | Sorafenib 200 mg (50-mg Tablet) | Sorafenib 400 mg (50-mg Tablet) | Sorafenib 400 mg (200-mg Tablet) | Sorafenib 400 mg (Expansion)
Serious Adverse Events (participants affected / at risk) | 5/7 | 1/3 | 8/12 | 9/17 | 76/119
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 11/12 | 16/17 | 118/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib 100 mg (50-mg Tablet) (N=7) | Sorafenib 200 mg (50-mg Tablet) (N=3) | Sorafenib 400 mg (50-mg Tablet) (N=12) | Sorafenib 400 mg (200-mg Tablet) (N=17) | Sorafenib 400 mg (Expansion) (N=119)
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 4
Platelets (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 6
Hemoglobin (HGB) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular arrhythmias (SVT/A FIB/FLUTT) (Cardiac disorders) | 0 | 0 | 0 | 1 | 4
Cardiovascular/arrhythmias - other (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coagulation - other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombosis/embolism (Cardiac disorders) | 0 | 0 | 1 | 3 | 8
Cardiac - ischemia/infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 3
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Pericardial effusion/pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 3
Phlebitis (superficial) (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Edema (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiovascular/general - other (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Dermatology/skin - other (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 10
Wound - infectious (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Wound - non-infectious (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Fever (in absence of neutropenia) (General disorders) | 0 | 0 | 0 | 1 | 7
Fatigue (Lethargy, Malaise, Asthenia) (General disorders) | 0 | 0 | 0 | 0 | 5
Constitutional symptoms - other (General disorders) | 0 | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 8
Dehydration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 8
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 6
Diarrhea, patients without colostomy (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Gastrointestinal - other (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3
Anorexia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia, esophagitis, odynophagia (painfull swallowing) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (radiographic or endoscopic) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Renal/genitourinary - other (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 4
Creatinine (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Ureteral obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
CNS Hemorrhage/belleding (Vascular disorders) | 0 | 0 | 2 | 0 | 1
Hemorrhage - other (Vascular disorders) | 0 | 0 | 0 | 0 | 3
Melena/GI bleeding (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hemoptysis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Rectal bleeding/hematochezia (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hemorrhage/bleeding with grade 3 or 4 thrombo (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hematuria (in absence of vaginal bleeding) (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Vaginal bleeding (Vascular disorders) | 0 | 0 | 0 | 0 | 1
SGPT (ALT) (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
SGOT (AST) (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (fever w/ unknow origin) (Infections and infestations) | 0 | 0 | 0 | 0 | 12
Infection without neutropenia (Infections and infestations) | 0 | 0 | 0 | 1 | 5
Infection (doc clinic or microbio) w/ GR 3 or 4 Neu (Infections and infestations) | 0 | 0 | 1 | 0 | 3
Infection with unknown ANC (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Infection/febrile neutropenia - other (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Amylase (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Lipase (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Neurology - other (Nervous system disorders) | 0 | 0 | 1 | 1 | 9
Syncope (fainting) (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Confusion (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Seizure(s) (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Ataxia (incoordination) (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Speech impairment (dysphasia or aphasia) (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy - motor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy - sensory (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pain - other (General disorders) | 0 | 0 | 0 | 1 | 10
Abdominal pain or cramping (General disorders) | 1 | 0 | 1 | 1 | 4
Chest pain (non-cardiac and nonpleuritic) (General disorders) | 1 | 0 | 0 | 0 | 3
Headache (General disorders) | 1 | 0 | 1 | 0 | 2
Tumor pain (onset/exacerb. tumor pain) (General disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 7
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib 100 mg (50-mg Tablet) (N=7) | Sorafenib 200 mg (50-mg Tablet) (N=3) | Sorafenib 400 mg (50-mg Tablet) (N=12) | Sorafenib 400 mg (200-mg Tablet) (N=17) | Sorafenib 400 mg (Expansion) (N=119)
Allergic reaction/hyper-sensitivity (Immune system disorders) | 3 | 0 | 0 | 5 | 20
Allergic rhinitis (Immune system disorders) | 0 | 0 | 0 | 0 | 12
Allergy/immunology - other (Immune system disorders) | 0 | 0 | 0 | 0 | 11
Auditory/hearing - other (Ear and labyrinth disorders) | 1 | 0 | 1 | 1 | 4
Inner ear/hearing (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Neutrophils/granolocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7 | 3 | 9 | 14 | 88
Platelets (Blood and lymphatic system disorders) | 2 | 3 | 8 | 11 | 77
Hemoglobin (HGB) (Blood and lymphatic system disorders) | 0 | 1 | 7 | 9 | 73
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2 | 36
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Edema (Cardiac disorders) | 0 | 1 | 3 | 1 | 24
Hypertension (Cardiac disorders) | 1 | 1 | 2 | 5 | 17
Thrombosis/embolism (Cardiac disorders) | 0 | 0 | 1 | 1 | 7
Phlebitis (superficial) (Cardiac disorders) | 0 | 0 | 0 | 1 | 5
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 1 | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 | 1 | 8 | 9 | 82
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 9 | 55
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1 | 6 | 6 | 47
Dermatology/skin - other (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 6 | 36
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 16
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 9
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 7
Wound - infectious (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 8
Flushing (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 5
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3
Bruising (in absence of GR 3 or 4 thrombo) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Fatigue (Lethargy, Malaise, Asthenia) (General disorders) | 7 | 1 | 6 | 9 | 97
Weight loss (General disorders) | 0 | 0 | 2 | 7 | 35
Fever (in absence of neutropenia) (General disorders) | 0 | 0 | 1 | 5 | 34
Constitutional symptoms - other (General disorders) | 1 | 1 | 0 | 4 | 27
Rigors, chills (General disorders) | 1 | 0 | 1 | 1 | 11
Sweating (diaphoresis) (General disorders) | 1 | 0 | 0 | 0 | 6
Nausea (Gastrointestinal disorders) | 6 | 2 | 6 | 8 | 78
Diarrhea, patients without colostomy (Gastrointestinal disorders) | 2 | 2 | 2 | 5 | 59
Anorexia (Gastrointestinal disorders) | 2 | 0 | 1 | 7 | 59
Vomiting (Gastrointestinal disorders) | 3 | 1 | 6 | 5 | 54
Constipation (Gastrointestinal disorders) | 5 | 1 | 2 | 4 | 33
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 0 | 0 | 3 | 5 | 29
Gastrointestinal - other (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 18
Dyspepsia/heartburn (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 16
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 11
Dehydration (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 9
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 7
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 5
Diarrhea, patients with colostomy (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 4
Ascites (non-malignant) (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Mouth dryness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Vascular disorders) | 0 | 0 | 3 | 2 | 25
Hemorrhage - other (Vascular disorders) | 0 | 0 | 0 | 1 | 10
Vaginal bleeding (Vascular disorders) | 1 | 0 | 0 | 0 | 0
SGOT (AST) (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 5
SGPT (ALT) (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 4
Bilirubin (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 4
Infection without neutropenia (Infections and infestations) | 3 | 0 | 5 | 9 | 44
Infection with unknown ANC (Infections and infestations) | 0 | 0 | 1 | 0 | 20
Infection/febrile neutropenia - other (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 28
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 9
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 11
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Lipase (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Metabolic/laboratory - other (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy - sensory (Nervous system disorders) | 6 | 2 | 5 | 9 | 73
Insomnia (Nervous system disorders) | 0 | 0 | 1 | 2 | 22
Mood alteration - depression (Nervous system disorders) | 0 | 0 | 0 | 4 | 21
Mood alteration - anxiety, agitation (Nervous system disorders) | 2 | 0 | 0 | 2 | 20
Neuropathy - motor (Nervous system disorders) | 1 | 0 | 1 | 1 | 20
Neurology - other (Nervous system disorders) | 0 | 0 | 1 | 1 | 14
Dizziness/lightheadedness (Nervous system disorders) | 0 | 0 | 0 | 1 | 13
Memory loss (Nervous system disorders) | 0 | 0 | 0 | 1 | 5
Confusion (Nervous system disorders) | 1 | 0 | 1 | 0 | 3
Syncope (fainting) (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Speech impairment (dysphasia or aphasia) (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Vision, blurred vision (Eye disorders) | 1 | 0 | 1 | 1 | 9
Ocular/visual - other (Eye disorders) | 0 | 0 | 1 | 1 | 4
Myalgia (muscle pain) (General disorders) | 2 | 0 | 4 | 8 | 65
Pain - other (General disorders) | 3 | 0 | 4 | 5 | 62
Arthralgia (joint pain) (General disorders) | 2 | 1 | 2 | 5 | 52
Abdominal pain or cramping (General disorders) | 1 | 1 | 3 | 3 | 29
Headache (General disorders) | 2 | 0 | 2 | 4 | 25
Bone pain (General disorders) | 1 | 1 | 1 | 1 | 17
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 2 | 0 | 0 | 0 | 15
Tumor pain (onset/exacerb. tumor pain) (General disorders) | 0 | 0 | 0 | 2 | 12
Neuropathic pain (jaw, neuro, limb pain) (General disorders) | 0 | 0 | 0 | 1 | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 6 | 56
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 5 | 37
Voice changes/stridor/larynx (hoarseness) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 16
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 9
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 4
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor recognizes right of principle investigator (PI) to publish results on completion of study, however, PI must provide draft of the communication to sponsor for approval 30 days prior to submission for publication. In case of difference of opinion between sponsor and PI, the parties will seek a solution satisfactory to both.